CLINICAL TRIAL: NCT00875888
Title: High Cut-off Continuous Venovenous Hemodialysis (CVVHD) to Improve Hemodynamic Stability and Organ Function Scores in Patients Treated for Acute Renal Failure After Systemic Inflammatory Response Syndrome (SIRS)/Septic Shock
Brief Title: High Cut-Off Continuous Veno-venous Hemodialysis (CVVHD) in Patients Treated for Acute Renal Failure After Systemic Inflammatory Response Syndrome (SIRS)/Septic Shock
Acronym: HICOSS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: based on interim analysis statistical significance in primary endpoint cannot be achieved with planned sample size, no safety concerns
Sponsor: Vantive Health LLC (Industry)
Collaborators: Gambro Dialysatoren GmbH (Industry); Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0000050; ISRCTN77656437
Record Dates: First submitted 2009-01-09; First posted 2009-04-06 (Estimated); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Systemic Inflammatory Response Syndrome; Kidney Failure, Acute
MeSH Terms: conditions — Systemic Inflammatory Response Syndrome; Acute Kidney Injury | interventions — Continuous Renal Replacement Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HCO (Experimental): High cut-off filters HCO1100
  Interventions: Device: continuous venovenous hemodialysis
- control (Active Comparator): conventional high-flux filters
  Interventions: Device: continuous venovenous hemodialysis

INTERVENTIONS:
Device: continuous venovenous hemodialysis — dialysate flow rate 35 ml/h/kg. Blood flow rate should be aimed at 200 ml/min, but not less than 150 ml/min. Bicarbonate- or lactate-buffered solutions will be used as dialysis fluids. Study dialyzers will be changed routinely every 24 h or earlier if the filter is obstructed by clotting.

SUMMARY:
This study will assess the influence of the High Cut-Off (HCO) CVVHD treatment on the disease progression in septic patients. The primary aim of the study is to evaluate whether HCO CVVHD leads to a significant improvement of the hemodynamic status (mean arterial pressure, vasopressor requirements) in septic patients in comparison to CVVHD treatment with conventional high-flux filters. For the HCO-group the investigators expect a 50% lower dosage of vasopressors needed to maintain an adequate organ perfusion.

DETAILED DESCRIPTION:
Severe sepsis is a devastating disorder that results from a complex host response to insult after infection. Despite advances in intensive care technologies sepsis remains an important and life-threatening problem. Sepsis is the most common cause of death in the intensive care unit.

Local or systemic release of bacteria-derived compounds, leading to the production of proinflammatory cytokines, induce systemic inflammatory reactions in septic patients. Continuous renal replacement therapies (CRRT) such as hemodialysis (CVVHD), hemofiltration (CVVH) or hemodiafiltration (CVVHDF) with conventional high-flux membranes allow to control fluid and electrolyte balance, and to improve the hemodynamic status of the patients. However, conventional high flux membranes have a limited permeability for sepsis-associated mediators with molecular weights in the range of 15.000 to 60.000 Da.

A promising approach to enhance the mediator removal is to use membranes having larger pores and permeability characteristics than those currently used in CRRT.

For that purpose a High Cut-Off (HCO) membrane has been developed and is manufactured by Gambro Research.After demonstrating the safety as well as the cytokine removal effectiveness in a clinical pilot study this study will assess the influence of the HCO treatment on the disease progression in septic patients.

ELIGIBILITY:
Inclusion Criteria:

1. Fulfilling at least two of the SIRS criteria as defined by the American College of Chest Physicians (ACCP)/Society of Critical Care Medicine (SCCM) Consensus Conference
2. Having signs of renal dysfunction
3. Requirement for catecholamine administration (norepinephrine or others)
4. Acute Physiology And Chronic Health Evaluation (APACHE II) score at enrolment greater than or equal to 19 and less than or equal to 30

Exclusion Criteria:

1. Lack of written informed consent from patients or a legally authorized surrogate
2. Duration of septic shock greater than 4 days
3. Hypoproteinemia (characterized by serum albumin less than 18 g/l)
4. End stage renal failure
5. Known active malignancy
6. Known human immunodeficiency virus (HIV), hepatitis B virus (HBV) or hepatitis C virus (HCV) infection
7. Age younger than 18 years or older than 80 years
8. Known pregnancy
9. Immunosuppression after transplantation
10. Participation in another clinical study
11. Renal replacement therapy greater than 24 hours before randomization

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2004-02; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Dosage of vasopressors | day 1 to day 5
Mean arterial pressure | day before inclusion and day 1 to day 5
Heart rate | day before inclusion and day 1 to day 5
Central venous pressure | day before inclusion and day 1 to day 5

SECONDARY OUTCOMES:
Sequential organ failure assessment (SOFA) score | at ICU admission, at inclusion and day 1 to day 5
Survival | 28 days
Length of need for catecholamine application | 28 days follow up
Length of need for mechanical ventilation | 28 days
Length of need for renal replacement therapy | 28 days
Length of stay in intensive care unit (ICU) | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Werner Beck, Dr., Study Director — Gambro Dialysatoren GmbH
Locations (4):
- Leopold Franzens Universität Innsbruck, Innsbruck, Austria
- Germany (3):
  - Medizinische Klinik mit Schwerpunkt Nephrologie Charite, Campus Mitte, Berlin
  - Charité-Virchow Klinik, Berlin
  - Universitätsklinikum Tübingen, Tübingen

REFERENCES:
- [Background] Morgera S, Haase M, Kuss T, Vargas-Hein O, Zuckermann-Becker H, Melzer C, Krieg H, Wegner B, Bellomo R, Neumayer HH. Pilot study on the effects of high cutoff hemofiltration on the need for norepinephrine in septic patients with acute renal failure. Crit Care Med. 2006 Aug;34(8):2099-104. doi: 10.1097/01.CCM.0000229147.50592.F9. PMID 16763508
- [Background] Morgera S, Haase M, Rocktaschel J, Bohler T, von Heymann C, Vargas-Hein O, Krausch D, Zuckermann-Becker H, Muller JM, Kox WJ, Neumayer HH. High permeability haemofiltration improves peripheral blood mononuclear cell proliferation in septic patients with acute renal failure. Nephrol Dial Transplant. 2003 Dec;18(12):2570-6. doi: 10.1093/ndt/gfg435. PMID 14605279
- [Background] Morgera S, Rocktaschel J, Haase M, Lehmann C, von Heymann C, Ziemer S, Priem F, Hocher B, Gohl H, Kox WJ, Buder HW, Neumayer HH. Intermittent high permeability hemofiltration in septic patients with acute renal failure. Intensive Care Med. 2003 Nov;29(11):1989-95. doi: 10.1007/s00134-003-2003-9. Epub 2003 Sep 3. PMID 12955174
- [Background] Morgera S, Haase M, Rocktaschel J, Bohler T, Vargas-Hein O, Melzer C, Krausch D, Kox WJ, Baumann G, Beck W, Gohl H, Neumayer HH. Intermittent high-permeability hemofiltration modulates inflammatory response in septic patients with multiorgan failure. Nephron Clin Pract. 2003;94(3):c75-80. doi: 10.1159/000072024. PMID 12902634
- [Background] Morgera S, Slowinski T, Melzer C, Sobottke V, Vargas-Hein O, Volk T, Zuckermann-Becker H, Wegner B, Muller JM, Baumann G, Kox WJ, Bellomo R, Neumayer HH. Renal replacement therapy with high-cutoff hemofilters: Impact of convection and diffusion on cytokine clearances and protein status. Am J Kidney Dis. 2004 Mar;43(3):444-53. doi: 10.1053/j.ajkd.2003.11.006. PMID 14981602